CLINICAL TRIAL: NCT04184401
Title: Effect of Albumin Administration Strategy for Ascites Replacement on Time to 1st Flatus After Liver Transplantation
Brief Title: Effect of Ascites Replacement Strategy on Time to 1st Flatus After LDLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: GC Pharma (Unknown)
Responsible Party: Principal Investigator, Ho Geol Ryu, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-1902-077-1011
Record Dates: First submitted 2019-11-12; First posted 2019-12-03 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Living Donor Liver Transplantation
Keywords: Ascites; Albumin; Hartmann's solution; Postoperative ileus
MeSH Terms: conditions — Ascites | interventions — Albumins; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Replacement with albumin (Experimental): 1. Check drain amount every 4 hour after SICU admission
  2. Replacement of 70% of drainage from previous 4 hours over next 4 hours
     * 30% of the drainage with 5% albumin
     * 40% of drainage with Hartmann's solution
     * If, serum K + level> 5mEq/L, replace with 0.9% saline instead of Hartmann solution
     * If, serum albumin level is below 2.6 g/dL, inject 100mL of 20% albumin
  Interventions: Drug: Ascites replacement with albumin and hartmann's solution
- Replacement with Hartmann's solution (Active Comparator): 1. Check drain amount every 4 hour after SICU admission
  2. Replacement of 70% of drainage from previous 4 hours with Hartmann's solution over next 4 hours
     * If, serum K + level> 5mEq/L, replace with 0.9% saline instead of Hartmann solution
     * If, serum albumin level is below 2.6 g/dL, inject 100mL of 20% albumin
  Interventions: Drug: Ascites replacement with hartmann's solution

INTERVENTIONS:
Drug: Ascites replacement with albumin and hartmann's solution — Combined strategy for ascites replacement
  * 30% of ascites: replacement with 5% albumin
  * 40% of ascites: replacement with Hartmann's solution
  Other Names: Experimental
  Arms: Replacement with albumin
Drug: Ascites replacement with hartmann's solution — Hartmann's solution only strategy for ascites replacement
  - 70% of ascites: replacement with Hartmann's solution
  Other Names: No intervention
  Arms: Replacement with Hartmann's solution

SUMMARY:
The aim of this study is to evaluate difference in the rate of recovery of intestinal motility according to different ascites replacement strategy after living donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (19 years or older)
* Elective living donor liver transplantation

Exclusion Criteria:

* Previous abdominal surgery
* Renal failure requiring renal replacement therapy
* Contraindications for 5% albumin use

  1. Condition with potential risk caused by increased circulating plasma (heart failure, renal failure combined with oliguria, pulmonary edema)
  2. Hemolytic anemia
* Contraindications for Hartmann solution

  1. Progressive lactic acidosis
  2. Hypervolemia
  3. Hypernatremia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Time to 1st flatus | within 4 weeks
  Interval between SICU admission and 1st flatus
Time to 1st diet | within 4 weeks
  Interval between SICU admission and 1st diet

CONTACTS AND LOCATIONS:
Overall Officials: Ho Geol Ryu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No